CLINICAL TRIAL: NCT01473550
Title: Mental Health Engagement Network (MHEN): Connecting Clients With Their Health Team
Brief Title: Mental Health Engagement Network (MHEN)
Acronym: MHEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other); Canadian Mental Health Association (Other); St. Joseph's Health Care London (Other)
Responsible Party: Principal Investigator, Cheryl Forchuk, Assistant Director, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 18451
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Mood Disorder; Psychotic Disorder
Keywords: Mental Health; Smart Technology; Mood disorder; Psychotic disorder
MeSH Terms: conditions — Mood Disorders; Psychotic Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Intervention (Experimental): At Phase 1 (first 3 months of project), the 200 participants in Group 1 will be provided with a Personal Health Record (PHR) through TELUS Health Space, as well as they will be introduced to smart phone technology to ready them for deployment of the prompts and reminders. Two months later, they will be provided with a smart phone.
  Interventions: Behavioral: Access to TELUS Health Space and Smart Phone
- Later Intervention (Experimental): A delayed implementation plan will be used (but will have no effect on the standard of care for the remaining 200 participants), so the remaining 200 participants in Group 2 will initially act as a control group, but at Phase 2 (six months later - approximately June 2012) the remaining 200 participants will be introduced to the technology in the same order (PHR -> Smart Phone). Group 2 will have the benefit of any enhancements made during Phase 1 of the project.
  Interventions: Behavioral: Access to TELUS Health Space and Smart Phone

INTERVENTIONS:
Behavioral: Access to TELUS Health Space and Smart Phone — Participants will be given their own TELUS Health Space and Smart Phone in order to have access to their personal health records. Specific procedures using the smart phone will depend on the individual care plan for each participant. Prompts and assessments will vary depending on participant needs.

SUMMARY:
Patients with mood disorder or psychotic disorder will be given handheld devices with personal health records to educate, monitor and deliver customizable healthcare tools based on their personal needs. The use of technology has great potential to deliver care more effectively and efficiently. No actual information is on the handheld device - it is accessed from a secure site behind hospital firewalls.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with mood disorder or psychotic disorder for a minimum one year
* Able to make informed consent to participate in the study
* Able to understand and speak English to the degree necessary to participate in interviews/focus groups

Exclusion Criteria:

* Younger than 18 or older than 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Lehman Quality of Life - Brief Version | Every 6 months for total of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Forchuk, PhD, Principal Investigator — Lawson Health Research Institute; University of Western Ontario
Locations (4):
- Canada (4):
  - Canadian Mental Health Association (London-Middlesex Branch), London, Ontario
  - Regional Mental Health Care, London, Ontario
  - London Health Sciences Centre, London, Ontario
  - Western Ontario Therapeutic Community Hostel, London, Ontario

REFERENCES:
- [Derived] Forchuk C, Donelle L, Ethridge P, Warner L. Client Perceptions of the Mental Health Engagement Network: A Secondary Analysis of an Intervention Using Smartphones and Desktop Devices for Individuals Experiencing Mood or Psychotic Disorders in Canada. JMIR Ment Health. 2015 Jan 21;2(1):e1. doi: 10.2196/mental.3926. eCollection 2015 Jan-Mar. PMID 26543906